CLINICAL TRIAL: NCT00121862
Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of the Leish-111f + MPL-SE Vaccine Compared to the Leish-111f Protein Alone in Montenegro Skin Test-Negative Healthy Adults
Brief Title: Study to Evaluate the Leish-111f + MPL-SE Vaccine in Healthy Adults Not Previously Exposed to Leishmania Parasite
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDRI-LCVPX-201
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2006-05

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmaniasis; Subunit Vaccine; Prevention; T cell
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis

INTERVENTIONS:
Biological: Leish-111f + MPL-SE vaccine

SUMMARY:
This study will evaluate the safety and immunogenicity of the Leish-111f + MPL-SE vaccine in adult subjects who have no evidence of previous exposure to the Leishmania parasite.

DETAILED DESCRIPTION:
Cutaneous leishmaniasis is a disfiguring disease that can progress to mucosal leishmaniasis, a more serious and possibly fatal form of Leishmania disease. All available medical therapies require weeks of treatment and cause significant toxicity.

It appears that Leishmania infections can be eliminated or prevented by T helper 1 immune responses. These findings argue that a vaccine that generates a T helper 1 response against the parasite will prevent the infection and disease. This is a phase 2, randomized, double blind, placebo-controlled study to evaluate the safety, tolerability and immunogenicity in Montenegro skin test (MST)-negative healthy adults of an investigational vaccine being developed for the prophylaxis of cutaneous leishmaniasis. The vaccine, identified as Leish-111f + MPL-SE, consists of a recombinant three-antigen Leishmania polyprotein (Leish-111f, 10 μg) together with the adjuvant MPL-SE (25 μg). In addition, the safety and immunogenicity of the vaccine will be compared to that of the Leish-111f protein (10 μg) given alone. The vaccine, Leish-111f protein alone or placebo will be given to each study subject three times at 4 week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Must have negative Montenegro skin test (0 mm)
* Must be in good general health with normal lab values
* Negative for HIV, hepatitis B and C

Exclusion Criteria:

* History of leishmaniasis or exposure to Leishmania vaccine or MPL-SE
* Nursing or pregnant female

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2005-08; Study Completion 2006-03

PRIMARY OUTCOMES:
Adverse events
Dose-limiting toxicities: hematology and serum chemistry evaluations at Screening, Days 7, 35, 63, 84
T-cell IFN-γ response to the Leish-111f protein: immunology evaluations at Days 0, 84, 168

SECONDARY OUTCOMES:
T-cell IL-5 response to the Leish-111f protein
Antibody responses to the Leish-111f protein
Skin test reactivity to the Leish-111f protein at Days 84, 168

CONTACTS AND LOCATIONS:
Overall Officials: Franco M Piazza, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Programa de Estudio y Control de Enfermedades Tropicales (PECET), Medellín, Colombia